CLINICAL TRIAL: NCT01505829
Title: Assessing Treatment Response of Peritoneal Metastases in Ovarian Cancer Using Diffusion Weighted Magnetic Resonance Imaging.
Brief Title: Diffusion-weighted Imaging Study in Cancer of the Ovary
Acronym: DISCOVAR
Status: Completed | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Cancer Research UK (Other); Royal Marsden NHS Foundation Trust (Other); Cambridge University Hospitals NHS Foundation Trust (Other); Imperial College Healthcare NHS Trust (Other); Northumbria Healthcare NHS Foundation Trust (Other); East and North Hertfordshire NHS Trust (Other Government)
Responsible Party: Principal Investigator, Nandita deSouza, Clinical Professor, Institute of Cancer Research, United Kingdom
Other Study IDs: 11/LO/1598 CCR3694; C1353/A12762 (Other Grant/Funding Number: Cancer Research UK)
Record Dates: First submitted 2011-11-18; First posted 2012-01-09 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Ovarian Cancer; Peritoneal Metastases
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour samples taken at surgery for histological analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Biological validation cohort 1
- Response assessment cohort 2

SUMMARY:
This project seeks to develop a quantitative imaging biomarker for evaluating and monitoring treatment response in ovarian cancer metastases and assess its potential in monitoring treatment response. This will involve standardising DW-MRI for the abdomen and pelvis across multiple centres and platforms, assessing reproducibility of the measurement in patients planned for neoadjuvant chemotherapy and assessing its utility as an early response biomarker in patients with platinum-sensitive relapse due to receive therapy with carboplatin. Scanning measurements will be correlated with histopathological markers in tumour samples in order to link the biomarker with response mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ovarian, primary peritoneal or fallopian tube cancer stage III or IV
* Scheduled to receive neoadjuvant chemotherapy (carboplatin/cisplatin)with planned debulking surgery.

Exclusion Criteria:

* Life expectancy of less than 6 months
* MRI contraindications
* Low grade or heavily calcified disease

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with primary or relapsed ovarian cancer
Sampling Method: Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-10-13 (Actual)

PRIMARY OUTCOMES:
Development of a Quantitative Imaging Biomarker for Evaluating Ovarian Cancer Metastases and Assessment of its Potential in Monitoring Treatment Response. | 4.0 years
  Diffusion-weighted magnetic resonance imaging (DW-MRI) for visualising peritoneal metastases will be developed.Reproducibility will be assessed in a multi-centre setting across multiple vendor platforms and field strengths by comparing 2 baseline scans per person and plotting absolute difference in ADC against mean of the 2 measurements.Biological validation will be achieved by correlating scan data (ADC change) following chemotherapy with histology of the tumour(amount of cell death) at surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Nandita deSouza, Professor, Principal Investigator — ICR
Locations (6):
- United Kingdom (6):
  - Addenbrookes Hospital, Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire
  - Queen Elizabeth Hospital, Newcastle, Gateshead
  - Mount Vernon Cancer Centre, Northwood, Middlesex
  - The Institute of Cancer Research and Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - Singleton Hospital, Swansea, Wales
  - Imperial College Healthcare NHS Trust, London

REFERENCES:
- [Derived] Winfield JM, Wakefield JC, Brenton JD, AbdulJabbar K, Savio A, Freeman S, Pace E, Lutchman-Singh K, Vroobel KM, Yuan Y, Banerjee S, Porta N, Ahmed Raza SE, deSouza NM. Biomarkers for site-specific response to neoadjuvant chemotherapy in epithelial ovarian cancer: relating MRI changes to tumour cell load and necrosis. Br J Cancer. 2021 Mar;124(6):1130-1137. doi: 10.1038/s41416-020-01217-5. Epub 2021 Jan 4. PMID 33398064